CLINICAL TRIAL: NCT07004322
Title: Investigation of Pharmacokinetics, Safety and Tolerability of Multiple Subcutaneous Doses of NNC0519-0130 in Male Chinese Participants With Overweight or Obesity
Brief Title: A Research Study of the New Medicine NNC0519-0130 in Male Chinese Participants Living With Excess Body Weight
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9541-4918; U1111-1283-0622 (Other: World Health Organization (WHO))
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus, Type 2; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NNC0519-0130 (Experimental): Participants will receive once weekly subcutaneous (s.c.) administration of NNC0519-0130 in dose escalation manner.
  Interventions: Drug: NNC0519-0130
- Placebo (Placebo Comparator): Participants will receive once weekly subcutaneous administration of placebo matched to NNC0519-0130.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NNC0519-0130 — NNC0519-0130 will be administered subcutaneously.
  Arms: NNC0519-0130
Drug: Placebo — Placebo matched to NNC0519-0130 will be administered subcutaneously.
  Arms: Placebo

SUMMARY:
Novo Nordisk is developing a new study medicine NNC0519-0130 to improve the treatment options for people living with type 2 diabetes and excess body weight. In this study, the concentration of NNC0519-0130 in the blood will be measured and its safety will be evaluated. The participants will either get NNC0519-0130 or placebo (a "dummy" substance), which treatment the participants get is decided by chance. This study will test up to 7 different doses of NNC0519-0130 and will last for about 28 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male Chinese participant.
* Body Mass Index (BMI) between 24.0 and 39.9 kilogram per square meter (kg/m^2) (both inclusive) at screening. Overweight should be due to excess adipose tissue, as judged by the investigator.
* Considered eligible based on the medical history, physical examination, and the results of vital signs, electrocardiogram (ECG) and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

* Any disorder which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol.
* Presence or history of any clinically relevant respiratory, metabolic, renal, hepatic, cardiovascular, gastrointestinal, or endocrinological conditions.
* Glycated haemoglobin (HbA1c) greater than or equal to (≥) 6.5 percentage (%) (48 millimoles per mole [mmol/mol]) at screening.
* Use of prescription medicinal products or non-prescription drugs (including Chinese traditional medicine or local medicine) within 14 days before screening, except routine vitamins, occasional use of paracetamol, ibuprofen, acetylsalicylic acid (ASA), domperidone or topical medication.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-26 (Actual); Primary Completion 2026-04-07 (Estimated); Study Completion 2026-04-07 (Estimated)

PRIMARY OUTCOMES:
AUC, NNC0519-0130, SS: Area under the NNC0519-0130 plasma concentration-time curve after the last dose in each treatment period | From pre-dose up to 7 days post-dose
  Measured in hours*nanomoles per liter (h*nmol/L).

SECONDARY OUTCOMES:
Cmax, NNC0519-0130, SS: Maximum plasma concentration of NNC0519-0130 after the last dose in each treatment period | From pre-dose up to 7 days post-dose
  Measured in nanomoles per liter (nmol/L).
t½, NNC0519-0130, SS: Terminal half-life of NNC0519-0130 after the last dose | From pre-dose until completion of the follow-up visit (day 162)
  Measured in hours (h).
Number of treatment emergent adverse events (TEAEs) | From time of first dosing (day 1) until completion of the end of study visit (day 162)
  Measured in number of events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Peking University Third Hospital, Northern Branch-Phase I, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com